CLINICAL TRIAL: NCT00714415
Title: Pharmacovigilance Evaluation Of Benefix (Registered) In Germany And Austria
Brief Title: Registry For Patients Treated With BeneFix In Usual Care Setting In Germany
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3090A1-4406; B1821011 (Other: Alias Study Number)
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with Hemophilia B
  Interventions: Drug: BeneFIX

INTERVENTIONS:
Drug: BeneFIX — Patients will be treated in accordance with the requirements of the labeling of BeneFIX in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.

SUMMARY:
The purpose of this observational study is to describe the incidence of adverse events among patients treated with BeneFix® in usual health care settings in Germany.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia B already receiving or starting treatment with reformulated BeneFIX®.

Exclusion Criteria:

* Patients with hemophilia B treated with a product other than BeneFIX®.
* Inclusion in the ongoing prospective registry of European hemophilia B patients using BeneFIX®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia B
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Allgemeines Krankenhaus Linz, Kinderklinik, Linz, Austria
- Germany (20):
  - Sonnengesundheitszentrum, München, Bavaria
  - Werlhof-Institut für Haemostaseologie GmbH, Hanover, Lower Saxony
  - Institut für Thrombophilie und Hämostaseologie, Münster, North Rhine-Westphalia
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Charite Campus Virchow-Klinikum, Padiatrie mit S. Hamatologie und Onkologie, Berlin
  - Kinder- und Jugendarzt-Praxis Blaubeuren, Blaubeuren Abbey
  - Institute of Experimental Haematology and Transfusion Medicine, Bonn
  - Praxis fur Kinder- und Jugendmedizin, Homoopathie, Brannenburg
  - Klinikum Bremen-Mitte gGmbH, Professor Hess Kinderklinik, Bremen
  - Gemeinschaftspraxis fuer Haematologie und Onkologie, Cologne
  - Klinikum Delmehorst gGmbH, Padiatrie, Delmenhorst
  - CRC Coagulation Research Centre GmbH, Duisburg
  - Universitaetsklinikum Duesseldorf, Klinik f. Kinder-Onkologie, Haematologie u. Klinische Immunologie, Düsseldorf
  - Klinikum der Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Eppendorf, Hamburg
  - SRH Kurpfalzkrankenhaus Heidelberg, Heidelberg
  - Klinikum Memmingen, Kinderklinik, Memmingen
  - Universitaetskinderklinik und Poliklinik im Dr. von Haunerschen, München
  - Universitaetsklinik fuer Kinder- und Jugendmedizin, Tübingen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090A1-4406&StudyName=Registry%20For%20Patients%20Treated%20With%20BeneFix%20In%20Usual%20Care%20Setting%20In%20Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- BeneFIX: On-Demand: Participants were treated with intravenous (IV) injection of BeneFIX whenever they had a bleeding episode, as a part of routine clinical practice at a dose and frequency prescribed by treating physician (with a mean recommended dose of 42.4 ± 16.6 international units per kilogram [IU/kg]). Participants were observed for up to a maximum duration of 8.7 years in this study.
- BeneFIX: Prophylaxis: Participants were treated prophylactically with a regular IV injection of BeneFIX to prevent any bleeding episode at a dose and frequency prescribed by treating physician (with a mean recommended dose of 34.4 ± 19.3 IU/kg). Participants were observed for up to a maximum duration of 8.7 years in this study.
Period: Overall Study
Arm/Group | BeneFIX: On-Demand | BeneFIX: Prophylaxis
Started | 25 | 55
Completed | 23 | 55
Not Completed | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix.
Groups:
- BeneFIX: On Demand: Participants were treated with IV injection of BeneFIX whenever they had a bleeding episode, as a part of routine clinical practice at a dose and frequency prescribed by treating physician (with a mean recommended dose of 42.4 ± 16.6 IU/kg). Participants were observed for up to a maximum duration of 8.7 years in this study.
- Total: Total of all reporting groups
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis | Total
Number analyzed (Participants) | 25 | 55 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.2 (18.8) | 16.0 (12.2) | 17.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 55 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; cancer; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to last visit (up to 8.7 years) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix.
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 25 | 55
participants
  AEs | 19 | 49
  SAEs | 8 | 29

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; cancer; congenital anomaly. AEs included both serious and non-serious. Relatedness to BeneFIX was assessed by the investigator.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix.
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 25 | 55
participants
  AEs | 2 | 8
  SAEs | 1 | 2

3. Primary Outcome: Number of Participants With Factor IX (FIX) Inhibitor Development as Measured by the Nijmegen-Modified Bethesda Assay
Description: FIX inhibitor development was defined as measured inhibitor titer of greater than (>) 0.6 Bethesda Units (BU) using the Nijmegen-modified Bethesda assay.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix.
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 25 | 55
participants | 1 | 3

4. Primary Outcome: Number of Participants With Adverse Events (AEs) of Special Interest
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Adverse Events of special interest included allergic reactions, less than expected therapeutic effect (LETE) of drug, lack of efficacy/low recovery, erythrocyte agglutination in tube or syringe red blood cell (RBC) agglutination phenomena and thrombogenicity.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix.
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 25 | 55
participants | 0 | 0

5. Primary Outcome: Investigator Assessment of Treatment Tolerability of Participants
Description: Investigator assessed the tolerability of participants and categorized as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: Safety analysis set included all participants with informed consent and treated with at least 1 dose of Benefix. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 23 | 54
participants
  Very good | 16 | 35
  Good | 7 | 18
  Moderate | 0 | 1
  Poor | 0 | 0

6. Primary Outcome: Participant Assessment of Treatment Tolerability
Description: Participants evaluated their treatment (BeneFIX) tolerability and rated it in 4 categories as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 22 | 52
participants
  Very good | 16 | 37
  Good | 6 | 14
  Moderate | 0 | 1
  Poor | 0 | 0

7. Secondary Outcome: Mean Total Number of Bleeding Episodes in Participants
Description: Participants documented all bleeding episodes in a diary during the study.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: Full analysis set included all participants with informed consent and treated with at least 1 dose of Benefix. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: bleeding episodes
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 22 | 54
bleeding episodes | 16.7 (21.2) | 17.6 (23.1)

8. Secondary Outcome: Mean Total Number of Bleeding Episodes Per Year in Participants
Description: Participants documented all bleeding episodes in a diary during the study. Mean total number of bleeding episodes per year was calculated by mean total number of bleeding episodes divided by duration of observation period (in years) for bleeding documentation.
Time Frame: Baseline until last visit (up to 8.7 years)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bleeding episodes per year
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 22 | 54
bleeding episodes per year | 4.7 (4.7) | 4.2 (4.3)

9. Secondary Outcome: Number of Participants With Change From Baseline Status in Number of Days Missed From School or Work
Description: Change from baseline status in days missed from school or work was categorized in 3 categories: Improvement, unchanged and worsening. Improvement was defined as a decrease in number of days missed by participants from school/work as compared to baseline; worsening was defined as an increase in number of days missed by participants from school/work as compared to baseline; unchanged was defined as no change in number of days missed by participants from school/work as compared to baseline. In this outcome measure, number of participants with change from baseline status (as improved, worsen, unchanged) in days missed from school/work were reported.
Time Frame: Baseline, up to 8.7 years
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 15 | 34
participants
  Improved | 4 | 7
  Unchanged | 9 | 20
  Worsened | 2 | 7

10. Secondary Outcome: Investigator Assessment of Treatment Efficacy of Participants
Description: Investigator evaluated the efficacy of BeneFIX in participants and rated it in 4 categories as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 23 | 54
participants
  Very good | 10 | 24
  Good | 11 | 30
  Moderate | 1 | 0
  Poor | 1 | 0

11. Secondary Outcome: Investigator Assessment of Treatment Handling of Participants
Description: Investigator evaluated the handling (administration) of BeneFIX by participants and rated it in 4 categories as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 23 | 54
participants
  Very good | 13 | 34
  Good | 10 | 20
  Moderate | 0 | 0
  Poor | 0 | 0

12. Secondary Outcome: Assessment of Treatment Efficacy by the Participants
Description: Participants evaluated the efficacy of BeneFIX and rated it in 4 categories as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 22 | 52
participants
  Very good | 11 | 27
  Good | 10 | 25
  Moderate | 0 | 0
  Poor | 1 | 0

13. Secondary Outcome: Assessment of Treatment Handling by the Participants
Description: Participants evaluated the handling (administration) of BeneFIX and rated it in 4 categories as very good, good, moderate and poor.
Time Frame: End of study visit (any time up to 8.7 years)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 22 | 52
participants
  Very good | 13 | 37
  Good | 8 | 15
  Moderate | 1 | 0
  Poor | 0 | 0

14. Secondary Outcome: Investigator Assessment of Treatment Satisfaction of Participants
Description: Investigator evaluated the participant's satisfaction of treatment with BeneFIX and rated it in 4 categories as very satisfied, satisfied, unsatisfied and very unsatisfied.
Time Frame: Baseline up to 8.7 years
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Number analyzed (Participants) | 23 | 54
participants
  Very satisfied | 12 | 27
  Satisfied | 9 | 27
  Unsatisfied | 1 | 0
  Very unsatisfied | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline until last visit (up to 8.7 years)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | BeneFIX: On Demand | BeneFIX: Prophylaxis
Serious Adverse Events (participants affected / at risk) | 8/25 | 29/55
Other Adverse Events (participants affected / at risk) | 18/25 | 46/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX: On Demand (N=25) | BeneFIX: Prophylaxis (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Middle ear disorder (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Dental cyst (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse event (General disorders) | 0 | 1
Complication associated with device (General disorders) | 0 | 1
Condition aggravated (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Mass (General disorders) | 0 | 1
Necrosis (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 3
Blister infected (Infections and infestations) | 0 | 1
Chronic tonsillitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Sports injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Angiogram (Investigations) | 0 | 1
Inhibiting antibodies positive (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Device defective (Product Issues) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar atrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arthrodesis (Surgical and medical procedures) | 0 | 1
Synovectomy (Surgical and medical procedures) | 0 | 1
Wisdom teeth removal (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX: On Demand (N=25) | BeneFIX: Prophylaxis (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Secondary hypogonadism (Endocrine disorders) | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 2 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Adverse event (General disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 4
Medical device discomfort (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Peripheral swelling (General disorders) | 0 | 3
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 3
Sensation of foreign body (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Allergy to venom (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Micrococcus infection (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 8
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 2
Accident at work (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 2 | 3
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 14
Face injury (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 7 | 21
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 3 | 5
Laceration (Injury, poisoning and procedural complications) | 3 | 10
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 12
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 7
Limb injury (Injury, poisoning and procedural complications) | 3 | 10
Lip injury (Injury, poisoning and procedural complications) | 0 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Mouth injury (Injury, poisoning and procedural complications) | 0 | 3
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1
Penis injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 7
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Sports injury (Injury, poisoning and procedural complications) | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Tongue injury (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 10
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 5 | 12
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Aspiration joint (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
CD4 lymphocytes decreased (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Oesophagoscopy (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 17
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 12
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 6
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 6
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 9
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Neuralgia (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1
Piriformis syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — This adverse event was reported in the participant who was the husband of woman who gave birth.
Device issue (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Renal failure (Renal and urinary disorders) | 0 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast haematoma (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Haemorrhage subepidermal (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Adenoidectomy (Surgical and medical procedures) | 1 | 0
Arthrodesis (Surgical and medical procedures) | 0 | 1
Artificial crown procedure (Surgical and medical procedures) | 1 | 0
Circumcision (Surgical and medical procedures) | 0 | 1
Dental care (Surgical and medical procedures) | 0 | 1
Ear tube insertion (Surgical and medical procedures) | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 0 | 1
Eye operation (Surgical and medical procedures) | 1 | 0
Gingivectomy (Surgical and medical procedures) | 1 | 0
Nail operation (Surgical and medical procedures) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 1 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 12
Haemorrhage (Vascular disorders) | 1 | 7
Hypertension (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures as primary and secondary was based on the study team's discretion, as it was not specified in source documents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.